CLINICAL TRIAL: NCT03718130
Title: A Phase 1, Randomized Trial to Assess the Safety, Reactogenicity, and Immunogenicity of a Combination HTNV and PUUV DNA Vaccine Candidate Administered by Electroporation
Brief Title: Combination HTNV and PUUV DNA Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); The Geneva Foundation (Other); US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency); Ichor Medical Systems Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-15-39
Record Dates: First submitted 2018-10-18; First posted 2018-10-24 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hantaan Virus Disease, Puumala Virus
MeSH Terms: conditions — Hantavirus Infections | interventions — tyramine-deoxysorbitol

STUDY DESIGN:
Intervention Model Description: 6 groups of 12 subjects each will receive varying vaccine dosages and vaccine candidate combinations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: 0.6 mg HTNV - Intradermal (ID) (Experimental): 0.1 mL 6.0 mg/mL HTNV DNA + 0.1 mL 0.9% saline (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Hantaan virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intradermal Delivery (ID)
- Group 2: 3.0 mg HTNV - Intramuscular (IM) (Experimental): 0.5 mL 6.0 mg/mL HTNV DNA + 0.5 mL 0.9% saline (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Hantaan virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intramuscular Delivery (IM)
- Group 3: 0.6 mg PUUV - Intradermal (ID) (Experimental): 0.1 mL 6.0 mg/mL PUUV DNA + 0.1 mL 0.9% saline (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID)
- Group 4: 3.0 mg PUUV - Intramuscular (IM) (Experimental): 0.5 mL 6.0 mg/mL PUUV DNA + 0.5 mL 0.9% saline (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intramuscular Delivery (IM)
- Group 5: 1.2 mg HTNV/PUUV (0.6 mg each) - Intradermal (ID) (Experimental): 0.1 mL 6.0 mg/mL HTNV DNA + 0.1 mL 6.0 mg/mL PUUV DNA (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Hantaan/Puumala (HTNV/PUUV) virus vaccines - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID)
- Group 6: 6.0 mg HTNV/PUUV (3.0 mg each) - Intramuscular (IM) (Experimental): 0.5 mL 6.0 mg/mL HTNV DNA + 0.5 mL 6.0 mg/mL PUUV DNA (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Interventions: Combination Product: Hantaan/Puumala (HTNV/PUUV virus vaccines - Using the TriGrid Delivery System (TDS) for Intramusular Delivery (IM)

INTERVENTIONS:
Combination Product: Hantaan virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intradermal Delivery (ID) — The HTNV vaccine will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: HTNV vaccine using TDS ID
  Arms: Group 1: 0.6 mg HTNV - Intradermal (ID)
Combination Product: Hantaan virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intramuscular Delivery (IM) — The HTNV vaccine will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: HTNV vaccine using TDS IM
  Arms: Group 2: 3.0 mg HTNV - Intramuscular (IM)
Combination Product: Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID) — The PUUV vaccine will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: PUUV vaccine using TDS ID
  Arms: Group 3: 0.6 mg PUUV - Intradermal (ID)
Combination Product: Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intramuscular Delivery (IM) — The PUUV DNA vaccine will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: PUUV vaccine using the TDS IM
  Arms: Group 4: 3.0 mg PUUV - Intramuscular (IM)
Combination Product: Hantaan/Puumala (HTNV/PUUV) virus vaccines - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID) — The HTNV and PUUV vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: HTNV/PUUV vaccines using the TDS ID
  Arms: Group 5: 1.2 mg HTNV/PUUV (0.6 mg each) - Intradermal (ID)
Combination Product: Hantaan/Puumala (HTNV/PUUV virus vaccines - Using the TriGrid Delivery System (TDS) for Intramusular Delivery (IM) — The HTNV and PUUV vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Other Names: HTNV/PUUV vaccines using the TDS IM
  Arms: Group 6: 6.0 mg HTNV/PUUV (3.0 mg each) - Intramuscular (IM)

SUMMARY:
To evaluate the safety and reactogenicity of the hantaan virus (HTNV), puumala virus (PUUV), and combination HTNV/PUUV DNA vaccine candidates delivered to healthy adults

DETAILED DESCRIPTION:
The development of DNA (deoxyribonucleic acid) vaccines, such as those to be utilized in this study, is based on the observation that antigen-encoding DNA plasmids can induce both cellular and humoral immune responses against various viral and bacterial pathogens. DNA vaccines are perceived as having a number of potential advantages over other types of vaccines. For example, DNA vaccines are easily constructed by recombinant technology; easily and inexpensively manufactured as a well-characterized molecule [DNA plasmid]; and at boost, not eliminated by prior immune response to the carrier or vector. Furthermore, as nonliving vaccines, they cannot lead to infection. The object of DNA vaccination is to deliver DNA into the nuclei of cells capable of presenting the encoded antigen to immune reactive cells that can elicit an immune response.

The study will enroll 6 randomized groups of 12 subjects each, for a total of 72 subjects. This approach will ensure at least 60 subjects complete all vaccinations at around 10 subjects per group, taking possible attrition into account. Subjects will receive one dose of vaccine on each of Days 0, 28, and 56 either intramuscularly or intradermally by electroporation and will be followed until Day 220.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or nonpregnant, nonlactating female, ages 18-49 (inclusive) at time of screening
* Have demonstrated adequate comprehension of the protocol by achieving a score of at least 80% correct on a short multiple-choice quiz. Individuals who fail to achieve a passing score on the initial quiz will be given the opportunity to retest after a review of the protocol information. Individuals who fail the quiz for the second time will not be enrolled.
* Have provided written informed consent before screening
* Subject is in good health as determined by past medical history, medication use, and abbreviated physical examination

  * Good health is defined by the absence of any medical condition described in the exclusion criteria in a subject with a normal abbreviated physical examination including vital signs. If the subject has another current, ongoing medical condition, the condition cannot meet any of the following criteria: (1) first diagnosed within 3 months of enrollment, (2) is worsening in terms of clinical outcome in last 6 months, or (3) involves need for medication that may pose a risk to subject's safety or impede assessment of adverse events or immunogenicity if they participate in the study.
  * An abbreviated physical examination differs from a complete physical examination in that it does not include a genitourinary and rectal examination.
* Available and able to participate for all study visits and procedures
* Sexually active men and women of childbearing potential must agree to use an effective method of contraception from 30 days prior to the first study vaccination until 6 months after the last study vaccination.

  * A sexually active man is defined as one whose partner is a woman of childbearing potential (see definition below) and has not had a vasectomy performed > 1 year prior to screening. They must agree not to father a child until 6 months after the last vaccination. These subjects must agree to use a barrier method of birth control (eg, either condom with spermicidal foam/gel/film/cream or partner usage of occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam/gel/film/cream/suppository).
  * Women of childbearing potential are defined as those who have not been sterilized via tubal ligation, bilateral oophorectomy, bilateral salpingectomy, hysterectomy, or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with history of documented radiological confirmation test at least 90 days after the procedure and are still menstruating or < 1 year of the last menses if perimenopausal. For this study, an effective contraceptive method is defined as one that results in a failure rate of less than 1% per year when it is used consistently and correctly (see the Manual of Procedures [MOP] for a list of acceptable methods).
* Female subjects agree to not donate eggs (ova, oocytes), and male subjects agree to not donate sperm from the start of screening until at least 6 months after the last vaccination.
* Negative hantavirus PsVNA test result at screening

Exclusion Criteria:

* History of prior infection with any hantavirus virus or prior participation in an HTNV, PUUV, or Andes virus vaccine trial.
* Has plans to travel to an area with endemic Hantaan, Puumala, Seoul, and Dobrava virus transmission during the study.

NOTE: Refer to the MOP for information on areas with endemic Hantaan, Puumala, Seoul, and Dobrava virus transmission

* History of severe local or systemic reactions to any vaccine or vaccine products or a history of severe allergic reactions.

  * This includes a known allergy to an aminoglycoside (eg, gentamicin, tobramycin, neomycin, and streptomycin).
* Is currently participating in or plans to participate in another study involving any investigational product (eg, vaccine, drug, or biologics) or a study that involves blood drawing, and/or an invasive procedure.

  * An invasive procedure includes endoscopy, bronchoscopy, or procedure requiring administration of IV contrast or removal of tissue.
* Receipt or planned receipt of any live vaccination, experimental or otherwise, within the period 30 days prior to or after each vaccination and receipt or planned receipt of an inactivated vaccination, experimental or otherwise, within the period of 14 days prior to or after each vaccination.
* Individuals, who based on clinical assessment by the investigator, have insufficient muscle mass to accommodate the 1 inch/25 mm penetration depth or have a skinfold thickness at eligible injection sites (deltoid region) that exceeds 40 mm.
* Individuals in whom the ability to observe local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Presence of any surgical or traumatic metal implants at the injection site (medial deltoid muscles or overlying skin).
* Screening laboratory results that are outside of the normal range (exceptions listed below) within 56 days prior to enrollment

  * Hemoglobin > 11.0 g/dL for women; > 12.9 g/dL for men
  * CBC (WBC and platelet) with differential either within institutional normal range or Grade 1 deviation from normal and deemed clinically insignificant
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.25x upper limit of normal (ULN)
  * Serum creatinine ≤ ULN
* Subjects with autoimmune disorders or chronic inflammatory disorders with a potential autoimmune correlation.
* Receipt of immunoglobulins and/or any blood products within the 120 days preceding screening or planned administration during the study period
* Donation of blood to a blood bank within 56 days prior to screening and at any time during the study period.
* Subject seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (anti-HCV).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, or use of anticancer chemotherapy or radiation therapy (cytotoxic) in the 3 years prior to screening.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Lyke, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 0.6 mg HTNV - Intradermal (ID): 0.1 mL 6.0 mg/mL HTNV DNA + 0.1 mL 0.9% saline (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantann virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intradermal Delivery (ID): The HTNV vaccine will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 2: 3.0 mg HTNV - Intramuscular (IM): 0.5 mL 6.0 mg/mL HTNV DNA + 0.5 mL 0.9% saline (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantann virus vaccine (HTNV) - Using TriGrid Delivery System (TDS) for Intramuscular Delivery (IM): The HTNV vaccine will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 3: 0.6 mg PUUV - Intradermal (ID): 0.1 mL 6.0 mg/mL PUUV DNA + 0.1 mL 0.9% saline (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID): The PUUV vaccine will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 4: 3.0 mg PUUV - Intramuscular (IM): 0.5 mL 6.0 mg/mL PUUV DNA + 0.5 mL 0.9% saline (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intramuscular Delivery (IM): The PUUV DNA vaccine will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID): 0.1 mL 6.0 mg/mL HTNV DNA + 0.1 mL 6.0 mg/mL PUUV DNA (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantaan/Puumala (HTNV/PUUV) virus vaccines - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID): The HTNV and PUUV vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM): 0.5 mL 6.0 mg/mL HTNV DNA + 0.5 mL 6.0 mg/mL PUUV DNA (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantaan/Puumala (HTNV/PUUV virus vaccines - Using the TriGrid Delivery System (TDS) for Intramusular Delivery (IM): The HTNV and PUUV vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
Period: Overall Study
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Started | 11 | 12 | 12 | 12 | 2 | 12
Completed | 0 | 11 | 0 | 12 | 0 | 12
Not Completed | 11 | 1 | 12 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM) | Total
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12 | 61
Age, Continuous [Mean (Full Range); unit: years] | 27.2 [22 to 41] | 33.3 [25 to 46] | 29.8 [22 to 43] | 37.2 [26 to 48] | 31.5 [29 to 34] | 28.6 [21 to 43] | 31.3 [21 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 9 | 1 | 9 | 44
  Male | 2 | 4 | 4 | 3 | 1 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 0 | 4 | 7
  Not Hispanic or Latino | 10 | 12 | 11 | 11 | 2 | 8 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 5 | 2 | 6 | 0 | 3 | 19
  Asian | 1 | 0 | 2 | 0 | 0 | 1 | 4
  White | 6 | 6 | 8 | 6 | 2 | 7 | 35
  Others | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Summary of Solicited Local Adverse Events (AEs)
Description: Summary of solicited local AEs occurring from the time of each injection through 14 days to evaluate the safety and reactogenicity of the HTNV, PUUV and combination HTNV/PUUV DNA vaccines
Time Frame: Days 0-14 after injection
Population: Summary of solicited local AE for Groups 1 through Group 6
Measure: Count of Participants; unit: Participants
Groups:
- Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM): 0.5 mL 6.0 mg/mL HTNV DNA + 0.5 mL 6.0 mg/mL PUUV DNA (IM) The HTNV and PUUV DNA vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantaan/Puumala (HTNV/PUUV virus vaccines - Using the TriGrid Delivery System (TDS) for Intramuscular Delivery (IM): The HTNV and PUUV vaccines will be administered using the IM TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12
Participants
  Dose 1 : Ecchymosis: None | 8 | 11 | 12 | 9 | 2 | 9
  Dose 1 : Ecchymosis: Mild | 3 | 0 | 0 | 2 | 0 | 2
  Dose 1 : Ecchymosis: Moderate | 0 | 1 | 0 | 1 | 0 | 1
  Dose 1 : Ecchymosis: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1 : Erythema: None | 6 | 11 | 6 | 12 | 1 | 9
  Dose 1 : Erythema: Mild | 2 | 1 | 1 | 0 | 1 | 1
  Dose 1 : Erythema: Moderate | 2 | 0 | 3 | 0 | 0 | 1
  Dose 1 : Erythema: Severe | 1 | 0 | 2 | 0 | 0 | 1
  Dose 1 : Induration (Hardness)/Swelling: None | 7 | 11 | 9 | 10 | 1 | 9
  Dose 1 : Induration (Hardness)/Swelling: Mild | 3 | 1 | 0 | 1 | 1 | 0
  Dose 1 : Induration (Hardness)/Swelling: Moderate | 0 | 0 | 2 | 1 | 0 | 1
  Dose 1 : Induration (Hardness)/Swelling: Severe | 1 | 0 | 1 | 0 | 0 | 2
  Dose 1 : Pain: None | 9 | 3 | 12 | 3 | 2 | 4
  Dose 1 : Pain: Mild | 2 | 8 | 0 | 8 | 0 | 6
  Dose 1 : Pain: Moderate | 0 | 1 | 0 | 1 | 0 | 2
  Dose 1 : Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1 : Tenderness: None | 4 | 4 | 7 | 3 | 1 | 5
  Dose 1 : Tenderness: Mild | 6 | 5 | 5 | 8 | 1 | 5
  Dose 1 : Tenderness: Moderate | 1 | 3 | 0 | 1 | 0 | 2
  Dose 1 : Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2 : Ecchymosis: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2 : Ecchymosis: None | 7 | 8 | 8 | 10 | 2 | 6
  Dose 2 : Ecchymosis: Mild | 0 | 1 | 0 | 0 | 0 | 1
  Dose 2 : Ecchymosis: Moderate | 1 | 2 | 0 | 2 | 0 | 0
  Dose 2 : Ecchymosis: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2 : Erythema: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2 : Erythema: None | 5 | 10 | 6 | 9 | 2 | 6
  Dose 2 : Erythema: Mild | 1 | 0 | 0 | 1 | 0 | 0
  Dose 2 : Erythema: Moderate | 1 | 1 | 1 | 1 | 0 | 1
  Dose 2 : Erythema: Severe | 1 | 0 | 1 | 1 | 0 | 0
  Dose 2 : Induration (Hardness)/Swelling: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2 : Induration (Hardness)/Swelling: None | 6 | 10 | 6 | 12 | 2 | 6
  Dose 2 : Induration (Hardness)/Swelling: Mild | 1 | 0 | 0 | 0 | 0 | 0
  Dose 2 : Induration (Hardness)/Swelling: Moderate | 0 | 1 | 2 | 0 | 0 | 1
  Dose 2 : Induration (Hardness)/Swelling: Severe | 1 | 0 | 0 | 0 | 0 | 0
  Dose 2 : Pain: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2 : Pain: None | 7 | 6 | 8 | 7 | 2 | 2
  Dose 2 : Pain: Mild | 0 | 5 | 0 | 4 | 0 | 5
  Dose 2 : Pain: Moderate | 1 | 0 | 0 | 1 | 0 | 0
  Dose 2 : Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2 : Tenderness: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2 : Tenderness: None | 5 | 5 | 7 | 4 | 2 | 2
  Dose 2 : Tenderness: Mild | 2 | 4 | 1 | 7 | 0 | 4
  Dose 2 : Tenderness: Moderate | 1 | 2 | 0 | 1 | 0 | 1
  Dose 2 : Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Ecchymosis: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3 : Ecchymosis: None | 3 | 9 | 4 | 11 | 2 | 2
  Dose 3 : Ecchymosis: Mild | 1 | 1 | 0 | 0 | 0 | 0
  Dose 3 : Ecchymosis: Moderate | 0 | 1 | 0 | 1 | 0 | 0
  Dose 3 : Ecchymosis: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Erythema: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3 : Erythema: None | 2 | 11 | 2 | 12 | 2 | 2
  Dose 3 : Erythema: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Erythema: Moderate | 1 | 0 | 1 | 0 | 0 | 0
  Dose 3 : Erythema: Severe | 1 | 0 | 1 | 0 | 0 | 0
  Dose 3 : Induration (Hardness)/Swelling: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3 : Induration (Hardness)/Swelling: None | 2 | 11 | 3 | 12 | 2 | 2
  Dose 3 : Induration (Hardness)/Swelling: Mild | 1 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Induration (Hardness)/Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Induration (Hardness)/Swelling: Severe | 1 | 0 | 1 | 0 | 0 | 0
  Dose 3 : Pain: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3 : Pain: None | 3 | 8 | 4 | 7 | 2 | 1
  Dose 3 : Pain: Mild | 0 | 3 | 0 | 5 | 0 | 1
  Dose 3 : Pain: Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Pain: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3 : Tenderness: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3 : Tenderness: None | 2 | 4 | 1 | 6 | 2 | 1
  Dose 3 : Tenderness: Mild | 1 | 6 | 2 | 6 | 0 | 1
  Dose 3 : Tenderness: Moderate | 1 | 1 | 1 | 0 | 0 | 0
  Dose 3 : Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Summary of Solicited Systemic Adverse Events (AEs)
Description: Summary of solicited systemic AEs occurring from the time of each injection through 14 days to evaluate the safety and reactogenicity of the HTNV, PUUV and combination HTNV/PUUV DNA vaccines
Time Frame: Days 0-14 after injection
Population: Summary of solicited systemic AE by Group and Dose Number, for Groups 1 through Group 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12
Participants
  Dose 1: Axillary Pain or Discomfort: None | 8 | 10 | 12 | 12 | 2 | 10
  Dose 1: Axillary Pain or Discomfort: Mild | 3 | 2 | 0 | 0 | 0 | 2
  Dose 1: Axillary Pain or Discomfort: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Axillary Pain or Discomfort: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Fatigue: None | 7 | 8 | 8 | 9 | 2 | 7
  Dose 1: Fatigue: Mild | 2 | 3 | 1 | 2 | 0 | 4
  Dose 1: Fatigue: Moderate | 1 | 1 | 3 | 1 | 0 | 1
  Dose 1: Fatigue: Severe | 1 | 0 | 0 | 0 | 0 | 0
  Dose 1: Headache: None | 7 | 10 | 10 | 10 | 2 | 9
  Dose 1: Headache: Mild | 3 | 1 | 0 | 1 | 0 | 2
  Dose 1: Headache: Moderate | 1 | 1 | 2 | 1 | 0 | 1
  Dose 1: Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Lymphadenopathy: None | 10 | 11 | 12 | 12 | 2 | 12
  Dose 1: Lymphadenopathy: Mild | 1 | 1 | 0 | 0 | 0 | 0
  Dose 1: Lymphadenopathy: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Lymphadenopathy: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Myalgia (Body aches/Muscular Pain): None | 10 | 6 | 11 | 9 | 2 | 7
  Dose 1: Myalgia (Body aches/Muscular Pain): Mild | 1 | 4 | 1 | 1 | 0 | 3
  Dose 1: Myalgia (Body aches/Muscular Pain): Moderate | 0 | 2 | 0 | 1 | 0 | 2
  Dose 1: Myalgia (Body aches/Muscular Pain): Severe | 0 | 0 | 0 | 1 | 0 | 0
  Dose 1: Tachypnea: None | 11 | 12 | 12 | 12 | 2 | 12
  Dose 1: Tachypnea: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Tachypnea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Tachypnea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Temperature: None | 11 | 11 | 12 | 11 | 2 | 12
  Dose 1: Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 1: Temperature: Moderate | 0 | 1 | 0 | 1 | 0 | 0
  Dose 1: Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Axillary Pain or Discomfort: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Axillary Pain or Discomfort: None | 6 | 11 | 8 | 10 | 2 | 7
  Dose 2: Axillary Pain or Discomfort: Mild | 1 | 0 | 0 | 2 | 0 | 0
  Dose 2: Axillary Pain or Discomfort: Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dose 2: Axillary Pain or Discomfort: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Fatigue: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Fatigue: None | 5 | 8 | 7 | 10 | 2 | 6
  Dose 2: Fatigue: Mild | 2 | 3 | 1 | 2 | 0 | 1
  Dose 2: Fatigue: Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dose 2: Fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Headache: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Headache: None | 4 | 9 | 7 | 11 | 2 | 7
  Dose 2: Headache: Mild | 4 | 1 | 1 | 1 | 0 | 0
  Dose 2: Headache: Moderate | 0 | 1 | 0 | 0 | 0 | 0
  Dose 2: Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Lymphadenopathy: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Lymphadenopathy: None | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Lymphadenopathy: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Lymphadenopathy: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Lymphadenopathy: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Myalgia (Body aches/Muscular pain): number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Myalgia (Body aches/Muscular pain): None | 8 | 7 | 8 | 9 | 2 | 5
  Dose 2: Myalgia (Body aches/Muscular pain): Mild | 0 | 4 | 0 | 2 | 0 | 1
  Dose 2: Myalgia (Body aches/Muscular pain): Moderate | 0 | 0 | 0 | 1 | 0 | 1
  Dose 2: Myalgia (Body aches/Muscular pain): Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Tachypnea: number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Tachypnea: None | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Tachypnea: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Tachypnea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Tachypnea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Temperature (fever): number analyzed (Participants) | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Temperature (fever): None | 8 | 11 | 8 | 12 | 2 | 7
  Dose 2: Temperature (fever): Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Temperature (fever): Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 2: Temperature (fever): Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Axillary pain or discomfort: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Axillary pain or discomfort: None | 3 | 11 | 4 | 12 | 2 | 2
  Dose 3: Axillary pain or discomfort: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Axillary pain or discomfort: Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Dose 3: Axillary pain or discomfort: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Fatigue: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Fatigue: None | 3 | 10 | 1 | 11 | 2 | 2
  Dose 3: Fatigue: Mild | 1 | 1 | 3 | 1 | 0 | 0
  Dose 3: Fatigue: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Headache: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Headache: None | 3 | 8 | 2 | 12 | 2 | 1
  Dose 3: Headache: Mild | 1 | 2 | 1 | 0 | 0 | 1
  Dose 3: Headache: Moderate | 0 | 1 | 1 | 0 | 0 | 0
  Dose 3: Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Lymphadenopathy: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Lymphadenopathy: None | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Lymphadenopathy: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Lymphadenopathy: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Lymphadenopathy: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Myalgia (Body aches/Muscular pain): number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Myalgia (Body aches/Muscular pain): None | 4 | 8 | 4 | 11 | 2 | 1
  Dose 3: Myalgia (Body aches/Muscular pain): Mild | 0 | 3 | 0 | 1 | 0 | 1
  Dose 3: Myalgia (Body aches/Muscular pain): Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Myalgia (Body aches/Muscular pain): Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Tachypnea: number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Tachypnea: None | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Tachypnea: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Tachypnea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Tachypnea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Temperature (fever): number analyzed (Participants) | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Temperature (fever): None | 4 | 11 | 4 | 12 | 2 | 2
  Dose 3: Temperature (fever): Mild | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Temperature (fever): Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Dose 3: Temperature (fever): Severe | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Subjects Experiencing Vaccine-related Unsolicited Adverse Events (AEs)
Description: Subjects experiencing vaccine-related unsolicited AEs from the time of the first injection through 28 days following each injection
Time Frame: Days 0-28 after injection
Population: Unsolicited Events that occurred across groups (Group 1 through Group 6) from the time of the first injection through 28 days following each injection
Measure: Count of Participants; unit: Participants
Groups:
- All Groups: Total Participants from Group 1 through 6
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM) | All Groups
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12 | 61
Participants
  Pruritus | 4 | 0 | 2 | 0 | 0 | 0 | 6
  Sore Throat | 0 | 1 | 0 | 1 | 0 | 1 | 3
  COVID-19 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Lightheadedness | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Muscle pain or spasms | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Viral illness/colds | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Back Pain | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Bacterial vaginitis | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Increased respiration | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Vomiting | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Ulcerative colitis | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Lump in armpit | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Constipation | 0 | 1 | 0 | 0 | 0 | 0 | 1
  AST elevation (Grade 3) | 0 | 0 | 1 | 0 | 0 | 0 | 1
  ALT elevation | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Seizure | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Scabbing | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Pus | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Influenza | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Nausea | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Fever | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Painful urination | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Nerve pain in limb | 0 | 0 | 0 | 0 | 0 | 1 | 1

4. Secondary Outcome: Proportion of Seropositive Subjects
Description: Determination of seropositive subjects (defined as PsVNA50 ≥ 1:20) at each scheduled time point
Time Frame: Days 0, 28, 56, 84, 140 and 220
Population: The planned enrolled sample size was 82 participants. A total of 61 participants were enrolled in the study. The reduction in total enrolled participants occurred due to the SARS-CoV-2 pandemic and study halt for ad Hoc Safety Monitoring Committee (SMC) review of an SAE required by the sponsor.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12
proportion of participants
  Day 0 | 0 [0 to 0.28] | 0 [0 to 0.26] | 0 [0 to 0.26] | 0 [0 to 0.26] | 0 [0 to 0.84] | 0.08 [0 to 0.38]
  Day 28: number analyzed (Participants) | 8 | 12 | 8 | 12 | 2 | 7
  Day 28 | 0.63 [0.24 to 0.91] | 0.42 [0.15 to 0.72] | 0.13 [0 to 0.53] | 0.08 [0 to 0.38] | 0 [0 to 0.84] | 0.14 [0 to 0.58]
  Day 56: number analyzed (Participants) | 3 | 12 | 5 | 12 | 2 | 2
  Day 56 | 0.67 [0.09 to 0.99] | 0.58 [0.28 to 0.85] | 0.4 [0.05 to 0.85] | 0.33 [0.1 to 0.65] | 0 [0 to 0.84] | 0.5 [0.01 to 0.99]
  Day 84: number analyzed (Participants) | 4 | 12 | 4 | 12 | 2 | 2
  Day 84 | 1 [0.4 to 1] | 0.75 [0.43 to 0.95] | 0.75 [0.19 to 0.99] | 0.33 [0.1 to 0.65] | 0 [0 to .84] | 0.5 [0.01 to 0.99]
  Day 140: number analyzed (Participants) | 11 | 12 | 11 | 12 | 2 | 0
  Day 140 | 0.73 [0.39 to 0.94] | 0.5 [0.21 to 0.79] | 0.09 [0 to 0.41] | 0.17 [0.02 to 0.48] | 0 [0 to 0.84] |
  Day 220: number analyzed (Participants) | 0 | 11 | 0 | 12 | 0 | 12
  Day 220 |  | 0.45 [0.17 to 0.77] |  | 0.08 [0 to 0.38] |  | 0.17 [0.02 to 0.48]

5. Secondary Outcome: Final Overall Rate of Seroconversion Over All Scheduled Time Points
Description: Determination of the final overall rate of serconversion over all scheduled time points to study completion for each study group. Seroconversion is defined as a post-vaccination HTNV- or PUUV-specific titer of ≥1:40, or a minimum four-fold rise compared to baseline titer, and all study volunteers will begin the study with a baseline titer <20 (ie, seronegative)
Time Frame: Days 0, 28, 56, 84, 140 and 220
Population: 1. Proportion of Seroconversion to HTNV PsVNA by Group and by Day
  2. Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12
proportion of participants
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 28: number analyzed (Participants) | 8 | 12 | 8 | 12 | 2 | 7
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 28 | 0.25 [0.03 to 0.65] | 0.25 [0.05 to 0.57] | 0 [0 to 0.37] | 0 [0 to 0.26] | 0 [0 to 0.84] | 0 [0 to 0.41]
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 56: number analyzed (Participants) | 3 | 12 | 5 | 12 | 2 | 2
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 56 | 0.33 [0.01 to 0.91] | 0.17 [0.02 to 0.48] | 0.2 [0.01 to 0.72] | 0.17 [0.02 to 0.48] | 0 [0 to 0.84] | 0 [0 to 0.84]
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 84: number analyzed (Participants) | 4 | 12 | 4 | 12 | 2 | 2
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 84 | 1 [0.4 to 1] | 0.5 [0.21 to 0.79] | 0 [0 to 0.6] | 0.08 [0 to 0.38] | 0 [0 to 0.84] | 0.5 [0.01 to 0.99]
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 140: number analyzed (Participants) | 11 | 12 | 11 | 12 | 2 | 12
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 140 | 0.27 [0.06 to 0.61] | 0.25 [0.05 to 0.57] | 0.09 [0 to 0.41] | 0.08 [0 to 0.38] | 0 [0 to 0.84] | 0 [0 to 0.26]
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 220: number analyzed (Participants) | 0 | 11 | 0 | 12 | 0 | 0
  Proportion of Seroconversion to HTNV PsVNA by Group and by Day: Day 220 |  | 0.09 [0 to 0.41] |  | 0 [0 to 0.26] |  |
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 28: number analyzed (Participants) | 8 | 12 | 8 | 12 | 2 | 7
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 28 | 0 [0 to 0.37] | 0 [0 to 0.26] | 0 [0 to 0.37] | 0.08 [0 to 0.38] | 0 [0 to 0.84] | 0 [0 to 0.41]
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 56: number analyzed (Participants) | 3 | 12 | 5 | 12 | 2 | 2
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 56 | 0 [0 to 0.71] | 0 [0 to 0.26] | 0 [0 to 0.52] | 0.33 [0.1 to 0.65] | 0 [0 to 0.84] | 0 [0 to 0.84]
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 84: number analyzed (Participants) | 4 | 12 | 4 | 12 | 2 | 2
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 84 | 0 [0 to 0.6] | 0.08 [0 to 0.38] | 0.75 [0.19 to 0.99] | 0.75 [0.43 to 0.95] | 0 [0 to 0.84] | 0 [0 to 0.84]
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 140: number analyzed (Participants) | 11 | 12 | 11 | 12 | 2 | 0
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 140 | 0 [0 to 0.28] | 0 [0 to 0.26] | 0.45 [0.17 to 0.77] | 0.42 [0.15 to 0.72] | 0 [0 to 0.84] |
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 220: number analyzed (Participants) | 0 | 11 | 0 | 12 | 0 | 12
  Proportion of Seroconversion to PUUV PsVNA80 by Group and by Day: Day 220 |  | 0 [0 to 0.28] |  | 0.17 [0.02 to 0.48] |  | 0 [0 to 0.26]

6. Secondary Outcome: Geometric Mean Titer (GMT) of the PsVNA50
Description: GMT of the PsVNA50 for HTNV- and PUUV-specific neutralizing antibodies at each schedule time point for each study group and over all time points for each study group
Time Frame: Days 0, 28, 56, 84, 140 and 220
Population: 1. Geometric Mean Titers of HTNV PsVNA80 by Group and by Day
  2. Geometric Mean Titers of PUUV PsVNA80 by Group and by Day
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
Number analyzed (Participants) | 11 | 12 | 12 | 12 | 2 | 12
titers
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 0 | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1]
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 28: number analyzed (Participants) | 8 | 12 | 8 | 12 | 2 | 7
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 28 | 28.68 [9.55 to 86.11] | 20.95 [13.28 to 33.06] | 14.1 [14.1 to 14.1] | 14.84 [13.26 to 16.6] | 14.1 [14.1 to 14.1] | 15.63 [12.15 to 20.11]
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 56: number analyzed (Participants) | 3 | 12 | 5 | 12 | 2 | 2
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 56 | 22.72 [2.92 to 177.01] | 22.06 [12.81 to 37.96] | 29.98 [5.81 to 154.64] | 17.35 [12.75 to 23.61] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1]
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 84: number analyzed (Participants) | 4 | 12 | 4 | 12 | 2 | 2
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 84 | 118.48 [17.97 to 781.08] | 42.65 [18.28 to 99.51] | 15.93 [10.8 to 23.52] | 17.53 [11.77 to 26.1] | 14.1 [14.1 to 14.1] | 24.91 [0.02 to 34375.75]
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 140: number analyzed (Participants) | 11 | 12 | 11 | 12 | 2 | 0
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 140 | 28.26 [14.98 to 53.32] | 22.7 [12.78 to 40.35] | 18.38 [10.18 to 33.16] | 15.93 [12.18 to 20.84] | 14.1 [14.1 to 14.1] |
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 220: number analyzed (Participants) | 0 | 11 | 0 | 12 | 0 | 12
  Geometric Mean Titers of HTNV PsVNA80 by Group and by Day: Day 220 |  | 15.5 [12.55 to 19.15] |  | 14.1 [14.1 to 14.1] |  | 14.58 [13.55 to 15.68]
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 0 | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1]
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 28: number analyzed (Participants) | 8 | 12 | 8 | 12 | 2 | 7
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 28 | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 22.36 [8.1 to 61.73] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1]
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 56: number analyzed (Participants) | 3 | 12 | 5 | 12 | 2 | 2
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 56 | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 15.27 [12.24 to 19.05] | 30.89 [13.86 to 68.82] | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1]
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 84: number analyzed (Participants) | 4 | 12 | 4 | 12 | 2 | 2
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 84 | 14.1 [14.1 to 14.1] | 17.7 [12.05 to 26.01] | 84.75 [12.33 to 582.34] | 69.97 [38.57 to 126.93] | 14.1 [14.1 to 14.1] | 21.57 [0.1 to 4786.68]
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 140: number analyzed (Participants) | 11 | 12 | 11 | 12 | 2 | 0
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 140 | 14.1 [14.1 to 14.1] | 14.1 [14.1 to 14.1] | 41.63 [20.39 to 84.97] | 31.54 [20.28 to 49.06] | 14.1 [14.1 to 14.1] |
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 220: number analyzed (Participants) | 0 | 11 | 0 | 12 | 0 | 12
  Geometric Mean Titers of PUUV PsVNA80 by Group and by Day: Day 220 |  | 14.1 [14.1 to 14.1] |  | 19.09 [13.12 to 27.77] |  | 14.1 [14.1 to 14.1]

ADVERSE EVENTS:
Time Frame: 6 months from last vaccination (Day 220)
Groups:
- Group 3: 0.6 mg PUUV - Intradermal (ID): 0.1 mL 6.0 mg/mL PUUV DNA + 0.1 mL 0.9% saline (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Puumala virus vaccine (PUUV) - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID): The PUUV vaccine will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
- Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID): 0.1 mL 6.0 mg/mL HTNV DNA + 0.1 mL 6.0 mg/mL PUUV DNA (ID) The HTNV and PUUV DNA vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroportation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
  Hantaan/Puumala (HTNV/PUUV) virus vaccines - Using the TriGrid Delivery System (TDS) for Intradermal Delivery (ID): The HTNV and PUUV vaccines will be administered using the ID TriGrid™ Delivery System (TDS), which utilizes the in vivo application of electrical fields (electroporation) to enhance the intracellular delivery of agents of interest in a targeted region of tissue.
Arm/Group | Group 1: 0.6 mg HTNV - Intradermal (ID) | Group 2: 3.0 mg HTNV - Intramuscular (IM) | Group 3: 0.6 mg PUUV - Intradermal (ID) | Group 4: 3.0 mg PUUV - Intramuscular (IM) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/12 | 0/2 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 1/12 | 0/12 | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 10/11 | 11/12 | 7/12 | 10/12 | 1/2 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 0.6 mg HTNV - Intradermal (ID) (N=11) | Group 2: 3.0 mg HTNV - Intramuscular (IM) (N=12) | Group 3: 0.6 mg PUUV - Intradermal (ID) (N=12) | Group 4: 3.0 mg PUUV - Intramuscular (IM) (N=12) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) (N=2) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM) (N=12)
ALT Elevation (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Alanine Aminotransferase Increased
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Generalized Tonic Clonic Seizure
Alcohol Withdrawal Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Alcoholic Seizure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: 0.6 mg HTNV - Intradermal (ID) (N=11) | Group 2: 3.0 mg HTNV - Intramuscular (IM) (N=12) | Group 3: 0.6 mg PUUV - Intradermal (ID) (N=12) | Group 4: 3.0 mg PUUV - Intramuscular (IM) (N=12) | Group 5: 1.2 mg HTNV/PUUV (0.6 mg Each) - Intradermal (ID) (N=2) | Group 6: 6.0 mg HTNV/PUUV (3.0 mg Each) - Intramuscular (IM) (N=12)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (11) | 1 (12) | 0 (0) | 3 (12) | 0 (0) | 3 (12) — Dose 1, Solicited Local AE
Erythema (Skin and subcutaneous tissue disorders) | 5 (11) | 1 (12) | 6 (12) | 0 (0) | 1 (2) | 3 (12) — Dose 1, Solicited Local AE
Induration (Hardness)/Swelling (General disorders) | 4 (11) | 1 (12) | 3 (12) | 2 (12) | 1 (2) | 3 (12) — Dose 1, Solicited Local AE
Pain (General disorders) | 2 (11) | 9 (12) | 0 (0) | 9 (12) | 0 (0) | 8 (12) — Dose 1, Solicited Local AE
Tenderness (General disorders) | 7 (11) | 8 (12) | 5 (12) | 9 (12) | 1 (2) | 7 (12) — Dose 1, Solicited Local AE
Ecchymosis (Skin and subcutaneous tissue disorders) | 1/8 (8) | 3/11 (11) | 0/8 (0) | 2 (12) | 0 (0) | 1/7 (7) — Dose 2, Solicited Local AE
Erythema (Skin and subcutaneous tissue disorders) | 3/8 (8) | 1/11 (11) | 2/8 (8) | 3 (12) | 0 (0) | 1/7 (7) — Dose 2, Solicited Local AE
Induration (Hardness)/Swelling (General disorders) | 2/8 (8) | 1/11 (11) | 2/8 (8) | 0 (0) | 0 (0) | 1/7 (7) — Dose 2, Solicited Local AE
Pain (General disorders) | 1/8 (8) | 5/11 (11) | 0/8 (0) | 5 (12) | 0 (0) | 5/7 (7) — Dose 2, Solicited Local AE
Tenderness (General disorders) | 3/8 (8) | 6/11 (11) | 1/8 (8) | 8 (12) | 0 (0) | 5/7 (7) — Dose 2, Solicited Local AE
Ecchymosis (Skin and subcutaneous tissue disorders) | 1/4 (4) | 2/11 (11) | 0/4 (0) | 1 (12) | 0 (0) | 0/2 (0) — Dose 3, Solicited Local AE
Erythema (Skin and subcutaneous tissue disorders) | 2/4 (4) | 0/11 (0) | 2/4 (4) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Local AE
Induration (Hardness)/Swelling (General disorders) | 2/4 (4) | 0/11 (0) | 1/4 (4) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Local AE
Pain (General disorders) | 1/4 (4) | 3/11 (11) | 0/4 (0) | 5 (12) | 0 (0) | 1/2 (2) — Dose 3, Solicited Local AE
Tenderness (General disorders) | 2/4 (4) | 7/11 (11) | 3/4 (4) | 6 (12) | 0 (0) | 1/2 (2) — Dose 3, Solicited Local AE
Axillary pain or discomfort (General disorders) | 3 (11) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 2 (12) — Dose 1, Solicited Systemic AE
Fatigue (General disorders) | 4 (11) | 4 (12) | 4 (12) | 3 (12) | 0 (0) | 5 (12) — Dose 1, Solicited Systemic AE
Headache (Nervous system disorders) | 4 (11) | 2 (12) | 2 (12) | 2 (12) | 0 (0) | 3 (12) — Dose 1, Solicited Systemic AE
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (11) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dose 1, Solicited Systemic AE
Myalgia (Body aches/Muscular pain) (Musculoskeletal and connective tissue disorders) | 1 (11) | 6 (12) | 1 (12) | 3 (12) | 0 (0) | 5 (12) — Dose 1, Solicited Systemic AE
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dose 1, Solicited Systemic AE
Temperature (fever) (General disorders) | 0 (0) | 1 (12) | 0 (0) | 1 (12) | 0 (0) | 0 (0) — Dose 1, Solicited Systemic AE
Axillary pain or discomfort (General disorders) | 2/8 (8) | 0/11 (0) | 0/8 (0) | 2 (12) | 0 (0) | 0/7 (0) — Dose 2, Solicited Systemic AE
Fatigue (General disorders) | 3/8 (8) | 3/11 (11) | 1/8 (8) | 2 (12) | 0 (0) | 1/7 (7) — Dose 2, Solicited Systemic AE
Headache (Nervous system disorders) | 4/8 (8) | 2/11 (11) | 1/8 (8) | 1 (12) | 0 (0) | 0/7 (0) — Dose 2, Solicited Systemic AE
Lymphadenopathy (Blood and lymphatic system disorders) | 0/8 (0) | 0/11 (0) | 0/8 (0) | 0 (0) | 0 (0) | 0/7 (0) — Dose 2, Solicited Systemic AE
Myalgia (Body aches/Muscular pain) (Musculoskeletal and connective tissue disorders) | 0/8 (0) | 4 (11) | 0/8 (0) | 3 (12) | 0 (0) | 2/7 (7) — Dose 2, Solicited Systemic AE
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0/8 (0) | 0/11 (0) | 0/8 (0) | 0 (0) | 0 (0) | 0/7 (0) — Dose 2, Solicited Systemic AE
Temperature (fever) (General disorders) | 0/8 (0) | 0/11 (0) | 0/8 (0) | 0 (0) | 0 (0) | 0/7 (0) — Dose 2, Solicited Systemic AE
Axillary pain or discomfort (General disorders) | 1/4 (4) | 0/11 (0) | 0/4 (0) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Systemic AE
Fatigue (General disorders) | 1/4 (4) | 1/11 (11) | 3/4 (4) | 1 (12) | 0 (0) | 0/2 (0) — Dose 3, Solicited Systemic AE
Headache (Nervous system disorders) | 1/4 (4) | 3/11 (11) | 2/4 (4) | 0 (0) | 0 (0) | 1/2 (2) — Dose 3, Solicited Systemic AE
Lymphadenopathy (Blood and lymphatic system disorders) | 0/4 (0) | 0/11 (0) | 0/4 (0) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Systemic AE
Myalgia (Body aches/Muscular pain) (Musculoskeletal and connective tissue disorders) | 0/4 (0) | 3/11 (11) | 0/4 (0) | 1 (12) | 0 (0) | 1/2 (2) — Dose 3, Solicited Systemic AE
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0/4 (0) | 0/11 (0) | 0/4 (0) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Systemic AE
Temperature (General disorders) | 0/4 (0) | 0/11 (0) | 0/4 (0) | 0 (0) | 0 (0) | 0/2 (0) — Dose 3, Solicited Systemic AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03718130/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03718130/SAP_001.pdf
  • Informed Consent Form (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03718130/ICF_002.pdf